CLINICAL TRIAL: NCT05631535
Title: Evaluation of the Efficacy of the Diabetes Prevention Program With a Very-low-energy Diet or a Low-energy Diet on Body Weight at 4 Months in Mexican Adults With Obesity: Two-armed-Randomized Controlled Trial
Brief Title: Obesity Treatment With a Very Low Energy Diet in Mexican Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Research Professor, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USO313008177
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Very Low Energy Diet
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with a very low-energy diet (Experimental)
  Interventions: Other: Intensive lifestyle change program with a very-low-energy diet
- Control group (Active Comparator)
  Interventions: Other: Intensive lifestyle change program with a low-energy diet

INTERVENTIONS:
Other: Intensive lifestyle change program with a very-low-energy diet — The intervention will consist of two phases. In the first phase, the participants receive weekly visits for two months. During these visits, a nutritionist will take the participants' weight and abdominal circumference measurements, and each one will receive a meal plan with a very low-energy diet (800 kcal/d). The second phase will implement in the third and fourth months, and nutritional counseling will continue to be provided every week in the third and biweekly in the fourth month. In this second phase, a gradual reintroduction to low-energy dietary meal plans (1200-1800 kcal/d) will perform. In addition, a specially adapted Diabetes Prevention Program for a very low-energy diet will implement.
  Arms: Intervention with a very low-energy diet
Other: Intensive lifestyle change program with a low-energy diet — The structure (frequency of nutritional counseling, number of sessions, time of sessions, etc.) in this group will be the same as that of the intervention group, and a modified Diabetes Prevention Program will also provide. From the beginning of the study will recommend meal plans with a low-energy diet (1200-1800 kcal).
  Arms: Control group

SUMMARY:
Clinical practice guidelines recommend behavioral change protocols for obesity treatment, such as the Diabetes Prevention Program, which involves a low-energy diet, physical activity recommendations, behavioral therapy, and frequent visits. Weight losses of 7-9% per year have achieve with this type of intervention. However, evidence suggests that a very low-energy diet may reach 10-15% weight loss and conduce superior clinical effects. Therefore, the objective will be to evaluate the efficacy of the Diabetes Prevention Program with a very-low energy diet and a low-energy diet on body weight change at four months in Mexican adults with obesity. The study will be a randomized controlled trial. Participants will be randomized to an intensive lifestyle change program with a very low-energy diet or an intensive lifestyle change program with a low-energy diet. The primary outcome will be a change in body weight. Secondary outcomes will be changes in waist circumference, body mass index, total body fat, fat-free mass, abdominal fat, blood pressure, and quality of life. Data will be analyzed on an intention-to-treat (ITT) using Student's t-tests or Mann-Whitney's U-test. The protocol was performed following the SPIRIT guidelines. Ethical approval was obtained from the Research Ethics Committee of the Department of Medicine of the University of Sonora.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 and ≤55 years of age).
* Residents of the city of Hermosillo, Sonora.
* BMI ≥ 30 and ≤ 40.
* Availability of time to participate in the study, including initial and final measurements.
* Have a device with access to the internet
* Availability and possibility to acquire the indicated diet
* Send a report of food consumption for three days

Exclusion Criteria:

* Being a participant in a weight loss program.
* Weight loss major than 5% in the last six months.
* Have type 2 diabetes or hypertension (previous).
* Use of drugs with an effect on body weight ( steroids, injectable progestins, lithium, valproic acid, carbamazepine, antipsychotics, antidepressants, thiazolidinediones, levothyroxine, metformin, and anorexigenic drugs).
* Have a history of coronavirus disease with hospitalization or the presence of sequelae that prevent the intervention from being carried out.
* Have cancer, kidney disease, eating disorders, psychiatric disorder (depression) or other serious diseases, active biliary disease, or known asymptomatic gallstones.
* Pregnancy or breastfeeding.
* Use of medications for obesity.
* Use of illegal substances harmful to health (drugs).
* Illiteracy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-06-02 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | Baseline to 16 weeks
  SECA medical body composition analyzer (mBCA) model 514 digital scale will be used. The participant should wear light clothing, remove footwear and metal objects, and have omitted food and beverages two hours before the measurement.

SECONDARY OUTCOMES:
Changes in body mass index | Baseline to 16 weeks
  It is necessary to divide the weight in kilograms by the height in centimeters squared.
Changes in waist circumference | Baseline to 16 weeks
  Participants will be measured standing at the umbilical level, using a Lufkin Executive anthropometric tape measure, model W606PMMX, from 0 to 200 cm.
Changes in body fat | Baseline to 16 weeks
  They will obtain it by Dual X-ray absorptiometry (DXA) with Quantitative Digital Radiography (QDR), Hologic Discovery A; Hologic, Inc. Bedford, Ma, USA.
Changes in fat-free mass | Baseline to 16 weeks
  They will obtain it by DXA with QDR, Hologic Discovery A; Hologic, Inc. Bedford, Ma, USA.
Changes in abdominal fat | Baseline to 16 weeks
  Estimation of abdominal fat, which includes visceral fat, will be obtained by DXA, QDR Hologic Discovery A; Hologic, Inc. Bedford, Ma, USA. For the definition of Region of Interest (ROI), will be used the APEX software version 3.0 and follow the criteria by the University of California (UCSF). The abdominal area will be selected as the ROI of the L2-upper iliac crest to monitor the change in abdominal fat. All body measurements will be taken in the dorsal decubitus position and at rest, without movement at the required time. If there is any movement during the measure, it will repeat with a limit of 2 attempts.
Changes in systolic blood pressure | Baseline to 16 weeks
  An Omron model HEM-907XL sphygmomanometer will be used to obtain the measurement in duplicate, following the methodology recommended by the American College of Cardiology (ACC) / American Heart Association (AHA).
Changes in diastolic blood pressure | Baseline to 16 weeks
  An Omron model HEM-907XL sphygmomanometer will be used to obtain the measurement in duplicate, following the methodology recommended by the American College of Cardiology (ACC) / American Heart Association (AHA).
Changes in perception of health-related quality of life | Baseline to 16 weeks
  The SF-36 Health Survey evaluates aspects of the quality of life in adult populations. This application generates eight concepts or scales of health, the result of the average of the sum of the points contains in the questionnaire for each item. These concepts are physical function, physical role, corporal pain, general health, vitality, social feature, emotional role, and mental health. The SF-36 is a self-applied instrument and contains 36 questions. For each scale, the answers to each question are coded and recoded (10 questions), and the results will be interprete on a scale of 0 to 100, the lowest results indicate poorer health, and the higher results are better health.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando G Díaz Zavala, Ph.D., Principal Investigator — Universidad de Sonora
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The data obtained will be available from the corresponding author on the research request.